CLINICAL TRIAL: NCT01705288
Title: Implementation of a Rapid Recovery Program in Gynecologic Oncology Surgery: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012LS096
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cervical Cancer; Uterine Endometrial Cancer; Ovarian Cancer
Keywords: laparotomy; hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms | interventions — Laparotomy; Morphine; Anesthesia, General; Anesthesia, Conduction; Anesthesia, Local; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Standard Laparotomy) (Active Comparator): Patients undergoing standard anesthesia and standard exploratory laparotomy. Treatment will be per your surgeon's routine standards.
  Interventions: Procedure: Laparotomy; Drug: intravenous narcotics; Drug: standard anesthesia
- Rapid Recovery Group (Experimental): Protocol for "rapid recovery laparotomy" procedure involves pre-operative counseling, the use of regional anesthesia (spinal or epidural pain management rather than intravenous narcotics), post-operative use of non-steroidal anti-inflammatory drugs, early eating after surgery, early walking, and certain goals for discharge from the hospital.
  Interventions: Procedure: Laparotomy; Drug: regional anesthesia; Drug: Non-steroidal anti-inflammatory drugs

INTERVENTIONS:
Procedure: Laparotomy — Exploratory surgery for gynecologic diagnosis.Involves pre-operative counseling, the use of regional anesthesia (spinal or epidural pain management rather than intravenous narcotics), early eating after surgery, early walking, and certain goals for discharge from the hospital
Drug: intravenous narcotics — given for pain management after surgery per physician orders
  Other Names: morphine
  Arms: Control Group (Standard Laparotomy)
Drug: standard anesthesia — inhalant or intravenous during surgery
  Other Names: general anesthesia
  Arms: Control Group (Standard Laparotomy)
Drug: regional anesthesia — given by spinal or epidural infusion
  Other Names: local anesthesia
  Arms: Rapid Recovery Group
Drug: Non-steroidal anti-inflammatory drugs — given for pain management after surgery
  Other Names: NSAIDs
  Arms: Rapid Recovery Group

SUMMARY:
Over 600,000 hysterectomies are performed annually in the United States. Despite increasing use of less invasive approaches, the majority of hysterectomies are still performed via traditional laparotomy, which can be associated with generally slower recovery and longer lengths of post-operative hospitalization. Rapid Recovery Protocols (RRP) seek to optimize post-surgical morbidity outcomes by returning a patient to normal physiology as quickly as possible following surgery.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to one of two groups: Rapid recovery protocol (regional anesthesia, pain control options with emphasis on nonsteroidal anti-inflammatory drugs (NSAIDS) over narcotic pain medications, early ambulation, and early enteral feeding) or standard of care (traditional laparatomy and supportive care).

ELIGIBILITY:
Inclusion Criteria:

* Women who are being seen at the Women's Health Center by the Gynecologic Oncology group at the University of Minnesota if planned surgery includes an exploratory laparotomy

Exclusion Criteria:

* < 19 years old
* Pregnant
* Undergoing a procedure other than laparotomy
* Scheduled to be discharged the same day of surgery
* Chronic narcotic pain medication user
* American Society of Anesthesiologists (ASA) score of > or = 3
* Any condition that would exclude women from undergoing regional anesthesia

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2016-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Argenta, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Chau JPC, Liu X, Lo SHS, Chien WT, Hui SK, Choi KC, Zhao J. Perioperative enhanced recovery programmes for women with gynaecological cancers. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD008239. doi: 10.1002/14651858.CD008239.pub5. PMID 35289396
- [Derived] Dickson EL, Stockwell E, Geller MA, Vogel RI, Mullany SA, Ghebre R, Witherhoff BJ, Downs LS Jr, Carson LF, Teoh D, Glasgow M, Gerber M, Rivard C, Erickson BK, Hutchins J, Argenta PA. Enhanced Recovery Program and Length of Stay After Laparotomy on a Gynecologic Oncology Service: A Randomized Controlled Trial. Obstet Gynecol. 2017 Feb;129(2):355-362. doi: 10.1097/AOG.0000000000001838. PMID 28079776

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group (Standard Laparotomy) | Rapid Recovery Group
Started | 52 | 51
Completed | 52 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (Standard Laparotomy) | Rapid Recovery Group | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 51 | 103
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 56.0 [52.8 to 59.2] | 55.4 [52.3 to 58.5] | 55.65 [52.8 to 58.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 103
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 51 | 103

OUTCOME MEASURES:

1. Primary Outcome: Hospital Stay
Description: Length of hospital stay for patients undergoing laparotomy on the gynecologic oncology service measured as whole days from the day of surgery until discharge
Time Frame: 1 Month
Population: Individuals randomized who underwent eligible surgery
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Control Group (Standard Laparotomy) | Rapid Recovery Group
Number analyzed (Participants) | 52 | 51
Days | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0]
Statistical Analysis 1: Comparison: Control Group (Standard Laparotomy) vs Rapid Recovery Group; Intention to Treat Analysis; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Medications Used
Description: Total daily narcotic pain medication used by patients. Narcotic use was standardized by conversion to morphine equivalents using the methods of Korff et al.
Time Frame: Post operative - day 2
Measure: Median (95% Confidence Interval); unit: Morphine equivalents
Arm/Group | Control Group (Standard Laparotomy) | Rapid Recovery Group
Number analyzed (Participants) | 51 | 48
Morphine equivalents | 10.0 [8.3 to 12.3] | 7.5 [3.3 to 10.0]
Statistical Analysis 1: Comparison: Control Group (Standard Laparotomy) vs Rapid Recovery Group; Intention to Treat Analysis; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pain Assessment
Description: Secondary outcome is to determine if rapid recovery can improve Visual Analogue Scale (VAS) for pain assessment. VAS scales are a horizontal line 100 mm in length with the left end labeled 'No pain' and the right end labeled 'Very severe pain'. The subject marks a point on the line that represents their perception of their current state. VAS score is determined by measuring the distance (mm) from the left end of the line to the point on the line marked by the subject. The range of possible values for this pain score is 0 to 100 mm.
Time Frame: Day 0
Population: Measured in early patients only
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | Control Group (Standard Laparotomy) | Rapid Recovery Group
Number analyzed (Participants) | 17 | 19
Score on a scale | 4.33 [3.0 to 6.25] | 3.13 [2.30 to 4.40]
Statistical Analysis 1: Comparison: Control Group (Standard Laparotomy) vs Rapid Recovery Group; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group (Standard Laparotomy) | Rapid Recovery Group
Serious Adverse Events (participants affected / at risk) | 1/52 | 4/51
Other Adverse Events (participants affected / at risk) | 4/52 | 7/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (Standard Laparotomy) (N=52) | Rapid Recovery Group (N=51)
ICU admission (General disorders) | 1 | 3 — The reason behind ICU admission is not recorded/details not available
Hemorrhage (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (Standard Laparotomy) (N=52) | Rapid Recovery Group (N=51)
Individual adverse events breakup not known (General disorders) | 4 | 7 — Only the counts of adverse events were available. The details of each adverse events data not available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes